CLINICAL TRIAL: NCT01476007
Title: Oral Versus Intramuscular Cobalamin to Treat Cobalamin Deficiency: Noninferiority Randomised Controlled Trial Pragmatic and Multi-center in the Primary Healthcare Setting (OB12 Project)
Brief Title: Oral/Intramuscular B12 to Treat Cobalamin Deficiency
Acronym: OB12
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gerencia de Atención Primaria, Madrid (Other Government)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Esperanza Escortell, Principal Investigator, Gerencia de Atención Primaria, Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010-024129-20; EC10-(115, 116, 117,119, 122) (Other Grant/Funding Number: Ministerio de Sanidad y Política Social)
Record Dates: First submitted 2011-11-15; First posted 2011-11-22 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Vitamin B 12 Deficiency
Keywords: primary health care; Vitamin B 12 Deficiency
MeSH Terms: conditions — Vitamin B 12 Deficiency | interventions — Vitamin B 12; Injections, Intramuscular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oral Cobalamin (vitamin B12) (Experimental): oral Cobalamin (vitamin B12)
  Interventions: Drug: oral Cobalamin (vitamin B12)
- intramuscular Cobalamin (vitamin B12) (Experimental): intramuscular Cobalamin (vitamin B12)
  Interventions: Drug: intramuscular Cobalamin (vitamin B12)

INTERVENTIONS:
Drug: oral Cobalamin (vitamin B12) — Intervention group: oral Optovite® B12 1000 gammas.
  Other Names: Optovite®
  Arms: oral Cobalamin (vitamin B12)
Drug: intramuscular Cobalamin (vitamin B12) — Control group: intramuscular Optovite® B12 1000 gammas.
  Other Names: Optovite® (intramuscular)
  Arms: intramuscular Cobalamin (vitamin B12)

SUMMARY:
Objective: To determine the effectiveness of oral versus intramuscular Cobalamin (vitamin B12) by restore cobalamin parameter in blood at 8, 26 and 52 weeks in ≥ 65 aged patients with Cobalamin Deficiency.

Design: Noninferiority randomised controlled trial, pragmatic and multi-center in the primary healthcare setting (Madrid Region).

Participants: ≥ 65 aged patients with Cobalamin Deficiency. Patients give inform consent. Number of patients: 320 (160 each arm). Assignment: randomized simple (automatic system).

Variables. Main outcome variable: Cobalamin level standardization (yes/no). Secondary outcome variables: Adverse events. Adherence measurement of treatment. Health related quality of life questionnaire (Euroqol-5D). Satisfaction and preferences. Other variables: Gender. Age. Live alone. Vegetarian diet. Alcohols consume. Clinic Variables (symptoms and physical examination) and blood parameters. Drugs consume.

Causes of all losses and withdrawals. Number of patients (age and gender) who declined to participate.

All data (excluding patient identification data) will be record in an electronic database.

Intervention group: oral Optovite® B12 1000 gammas. Control group: idem intramuscular.

Analysis: Descriptive analysis (screening phase). Baseline comparison of the two intervention groups. Effect of cobalamin (main outcome variable). Security. Quality of life. Adherence measurement of treatment.

DETAILED DESCRIPTION:
Variables. Main outcome variable: Cobalamin level standardization (yes/no). Secondary outcome variables: Adverse events. Adherence measurement of treatment. Health related quality of life questionnaire (Euroqol-5D). Satisfaction and preferences. Other variables: Gender. Age. Live alone. Vegetarian diet. Alcohols consume. Clinic Variables (symptoms and physical examination) and blood parameters. Drugs consume.

Causes of all losses and withdrawals. Number of patients (age and gender) who declined to participate.

All data (excluding patient identification data) will be record in an electronic database.

Intervention group: oral Optovite® B12 1000 gammas. Control group: idem intramuscular.

Analysis: Descriptive analysis (screening phase). Baseline comparison of the two intervention groups. Effect of cobalamin (main outcome variable). Security. Quality of life. Adherence measurement of treatment.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 65 aged patients with Cobalamin Deficiency.
* Patients give inform consent.

Exclusion Criteria:

* Treatment with B12 (1 last year)
* Neurologic or psychiatric pathologies
* Folic acid < 2.3ng/ml ...

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 284 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
Change from Cobalamin level standardization | 1 year
  Change from Baseline in Cobalamin level at 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rosario Riesgo, MD, Principal Investigator — Gerencia Atención Primaria. Madrid; Teresa Sanz-Cuesta, MD, Study Director — Gerencia Atención Primaria. Madrid; Isabel DelCura-González, MD Phd, Principal Investigator — Gerencia Atención Primaria. Madrid; Jesús Martín-Fernández, MD Phd, Principal Investigator — Gerencia Atención Primaria. Madrid; Sofía Garrido-Elustondo, MD, Principal Investigator — Gerencia Atención Primaria. Madrid; Esperanza Escortell-Mayor, MD Phd, Principal Investigator — Gerencia Atención Primaria. Madrid
Locations (1):
- Gerencia Atención Primaria, Madrid, Madrid, Spain

REFERENCES:
- [Background] Sanz-Cuesta T, Gonzalez-Escobar P, Riesgo-Fuertes R, Garrido-Elustondo S, del Cura-Gonzalez I, Martin-Fernandez J, Escortell-Mayor E, Rodriguez-Salvanes F, Garcia-Solano M, Gonzalez-Gonzalez R, Martin-de la Sierra-San Agustin MA, Olmedo-Luceron C, Sevillano Palmero ML, Mateo-Ruiz C, Medina-Bustillo B, Valdivia-Perez A, Garcia-de Blas-Gonzalez F, Marino-Suarez JE, Rodriguez-Barrientos R, Ariza-Cardiel G, Cabello-Ballesteros LM, Polentinos-Castro E, Rico-Blazquez M, Rodriguez-Monje MT, Soto-Diaz S, Martin-Iglesias S, Rodriguez-Gonzalez R, Breton-Lesmes I, Vicente-Herrero M, Sanchez-Diaz J, Gomez-Gascon T, Drake-Canela M, Asunsolo-del Barco A; OB12 Group. Oral versus intramuscular administration of vitamin B12 for the treatment of patients with vitamin B12 deficiency: a pragmatic, randomised, multicentre, non-inferiority clinical trial undertaken in the primary healthcare setting (Project OB12). BMC Public Health. 2012 May 31;12:394. doi: 10.1186/1471-2458-12-394. PMID 22650964
- [Derived] Sanz-Cuesta T, Escortell-Mayor E, Cura-Gonzalez I, Martin-Fernandez J, Riesgo-Fuertes R, Garrido-Elustondo S, Marino-Suarez JE, Alvarez-Villalba M, Gomez-Gascon T, Gonzalez-Garcia I, Gonzalez-Escobar P, Vargas-Machuca Cabanero C, Noguerol-Alvarez M, Garcia de Blas-Gonzalez F, Banos-Morras R, Diaz-Laso C, Caballero-Ramirez N, Herrero de-Dios A, Fernandez-Garcia R, Herrero-Hernandez J, Pose-Garcia B, Sevillano-Palmero ML, Mateo-Ruiz C, Medina-Bustillo B, Aguilar-Jimenez M; OB12 Group. Oral versus intramuscular administration of vitamin B12 for vitamin B12 deficiency in primary care: a pragmatic, randomised, non-inferiority clinical trial (OB12). BMJ Open. 2020 Aug 20;10(8):e033687. doi: 10.1136/bmjopen-2019-033687. PMID 32819927